CLINICAL TRIAL: NCT04546919
Title: the Mechanism of the Downregulation of R-spondin3 in Sepsis Induced Lung Injury
Brief Title: Effect of R-spondin3 on Sepsis Induced Endothelial Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XHEC-C-2020-084
Record Dates: First submitted 2020-08-19; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-07

CONDITIONS: Acute Lung Injury (ALI); Acute Respiratory Distress Syndrome (ARDS)
Keywords: sepsis; Rspondin3; ALI
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood samples from septic patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sepsis — Body temperature higher than 38°C or lower than 36°C; Heart rate higher than 90/min; Hyperventilation evidenced by respiratory rate higher than 20/min or PaCO2 lower than 32 mmHg; White blood cell count higher than 12,000 cells/ µl or lower than 4,000/ µl.

SUMMARY:
Sepsis is the most frequent risk factor for ALI/ARDS. Meanwhile, Pulmonary is the most vulnerable organ to fail in response to sepsis, vascular endothelial dysfunction is a central event in the pathophysiology of sepsis. An improved understanding of endothelial response and associated biomarkers may lead to strategies to more accurately predict outcome and develop novel endothelium-directed therapies in sepsis.

The human and mouse R-spondins encode a family of proteins that includes four paralogs (R-spo1-4). R-spondins are secreted proteins found primarily in the extracellular region and are known to promote β-catenin signaling. Among them, the embryonic lethal vascular remodeling phenotype of R-spondin3 (Rspo3) mutant mice suggests a role of EC derived Rspo3 in angiogenesis. Rspo3 protects tissues against mesenteric I/R by tightening endothelial cell junction and improving vascular intergrity. However, the role of Rspo3 in sepsis-induced pulmonary endothelial dysfunction remains unclear. Thus, it is worthwhile to explore the relationship between Rspo3 and sepsis-induced lung injury, which will be helpful for prevention and treatment of sepsis-induced lung injury and endothelial dysfunction.

DETAILED DESCRIPTION:
Acute lung injury (ALI) or acute respiratory distress syndrome (ARDS), is a clinical problem induced by acute and excessive pulmonary inflammation. Sepsis is the most frequent risk factor for ALI/ARDS. Meanwhile, Pulmonary is the most vulnerable organ to fail in response to sepsis, and a major cause of death for sepsis patients is respiratory failure. Despite modern clinical practices in critical care medicine, there still remains a mortality rate as high as 45%. In addition, Vascular endothelial dysfunction is a central event in the pathophysiology of sepsis. Endothelial cell activation is associated with sepsis severity, organ dysfunction and mortality. An improved understanding of endothelial response and associated biomarkers may lead to strategies to more accurately predict outcome and develop novel endothelium-directed therapies in sepsis.

The human and mouse R-spondins encode a family of proteins that includes four paralogs (R-spo1-4). R-spondins are secreted proteins found primarily in the extracellular region and are known to promote β-catenin signaling. Among them, the embryonic lethal vascular remodeling phenotype of R-spondin3 (Rspo3) mutant mice suggests a role of EC derived Rspo3 in angiogenesis. Former studies demonstrated that endothelial Rspo3 enhances cell autonomous non-canonical Wnt signaling, thereby preventing retinal and tumor blood vessel regression and EC apoptosis. The mid-gestational lethality of Rspo3-ECKO mice indicated a role of EC-derived RSPO3 in controlling blood vessel remodeling. Furthermore, Rspo3 protects tissues against mesenteric I/R by tightening endothelial cell junction and improving vascular intergrity. However, the role of Rspo3 in sepsis-induced pulmonary endothelial dysfunction remains unclear. Thus, it is worthwhile to explore the relationship between Rspo3 and sepsis-induced lung injury.

In the present study, the investigators will analyze the expression of Rspo3 in septic patients and sepsis-induced lung injury models and explore whether Rspo3 could protect sepsis-associated lung injury, which will be helpful for prevention and treatment of sepsis-induced lung injury and endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* patients with sepsis defined as SIRS combined with an infectious episode and dysfunction of one or more organ
* age older than 18 years

SIRS is considered to be present when patients have more than one of the following clinical findings:

* Body temperature higher than 38°C or lower than 36°C;
* Heart rate higher than 90/min
* Hyperventilation evidenced by respiratory rate higher than 20/min or PaCO2 lower than 32 mmHg;
* White blood cell count higher than 12,000 cells/ µl or lower than 4,000/ µl.

Exclusion Criteria:

* patients younger than 18
* women during pregnancy or lactation; being involved in other clinical subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: septic patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-08-08 (Estimated); Study Completion 2021-12-12 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma Concentration of R-spondin 3 | after initiation of sepsis within 24 hours
  The venous blood samples were collected from septic patients after the onset of the sepsis, plasma were separated by centrifugation and detected for R-spondin3 concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Jiang, chief doctor, Study Chair — Xinhua Hospital affiliated to Medicine school,Shanghai Jiaotong University
Locations (1):
- Department of Anesthesia, Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT04546919/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT04546919/ICF_001.pdf